CLINICAL TRIAL: NCT06518382
Title: A Retrospective Observational Study Characterizing Tumour-microenvironment Spatial Interaction Aimed at the Identification of New Markers of Resistance to Therapy in HER2-positive Breast Cancer Patients
Brief Title: Tumor-microenvironment Spatial Interaction to Identify Markers of Resistance to Therapy in HER2+ Breast Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Giampaolo Bianchini (Other)
Responsible Party: Sponsor-Investigator, Giampaolo Bianchini, Head of Breast Cancer Group, Department of Medical Oncology -PI-, IRCCS Ospedale San Raffaele
Organization: IRCCS Ospedale San Raffaele (Other)
Other Study IDs: TaME-HER2BrCa
Record Dates: First submitted 2024-07-16; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective observational study aims at the comparison of the tumour-microenvironment tissue architecture before and after neo-adjuvant therapy in samples from HER2-positive (HER2+) breast cancer (BrCa) patients that display residual invasive disease in the breast/lymph node at surgery after standard-of-care combined chemotherapy and trastuzumab treatment.

The working hypothesis of the investigators is that:

Therapy imposes a selective pressure on tumour-microenvironment features promoting resistance to treatment.

Participant that have already undergone neo-adjuvant treatment as part of their regular medical care for HER2-positive breast cancer will provide access to formalin-fixed paraffin-embedded (FFPE) samples taken before and after therapy.

Tumoral, peri-tumoral and stromal regions of each specimen will be analyzed with the ultimate goal to identify new biomarkers (and putative targets) of resistance to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation in the study.
2. Patient underwent the following procedure before surgery: biopsy, sequential chemotherapy comprising treatment with antracyclines (AC/EC q21, 4 cycles) followed by taxanes (paclitaxel 1,8,15 q21 for 12 weeks) in combination with the anti-HER2 antibody trastuzumab.
3. Specimen collected at surgery display residual invasive disease in the breast/lymph node.

Exclusion Criteria:

1. pre-existing conditions or concurrent diagnoses;
2. concomitant use of other medications during neo-adjuvant treatment;
3. quality of stored specimen does not meet the standard for Imaging Mass Cytometry analysis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2+ Breast Cancer patients displaying residual invasive disease in the breast/lymph node at surgery after neo-adjuvant treatment [sequential chemotherapy comprising treatment with antracyclines (AC/EC q21, 4 cycles) followed by taxanes (paclitaxel 1,8,15 q21 for 12 weeks) in combination with the anti-HER2 antibody trastuzumab].
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
number of different cells per each phenotype | before and within 3 months from neo-adjuvant therapy (at surgery)
  Cell types will be classified based on the expression of specific lineage/phenotype markers.
density of each phenotype | before and within 3 months from neo-adjuvant therapy (at surgery)
  Cell phenotype densities will be calculated by dividing the number of total cells counted by the total area of the tissue acquired.
fraction of proliferative/active cells of each phenotype | before and within 3 months from neo-adjuvant therapy (at surgery)
  The proportion of cells positive for the proliferation marker Ki67 will be assessed per cell phenotype. To assess the proportion of active immune cells, we will quantify the expression level of activation markers.
frequency of interactions | before and within 3 months from neo-adjuvant therapy (at surgery)
  Cells will be defined as partaking in an interaction if their whole-cell profiles are in direct contact (contiguous pixels). Cell phenotypes will be mapped to cell-cell interaction masks, and for each specimen proximity events (cell-cell interactions) will be classified as homotypic or heterotypic proximity events
frequency of functional crosstalk events | before and within 3 months from neo-adjuvant therapy (at surgery)
  Cells will be defined as participating in a functional crosstalk event if the proximal (contiguous pixels) cells express functional pairs (receptor/ligand) of markers (e.g. PD1/PDL1).
  The frequency of functional crosstalk events will be computed as the number of interactions between cells expressing functional pairs divided by the total number of cells expressing one of the markers (receptor, e.g. PD1) in the specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Giampaolo Bianchini, MD, Principal Investigator — Head Breast Cancer Group - Department of Medical Oncology - IRCCS San Raffaele Hospital
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang XQ, Danenberg E, Huang CS, Egle D, Callari M, Bermejo B, Dugo M, Zamagni C, Thill M, Anton A, Zambelli S, Russo S, Ciruelos EM, Greil R, Gyorffy B, Semiglazov V, Colleoni M, Kelly CM, Mariani G, Del Mastro L, Biasi O, Seitz RS, Valagussa P, Viale G, Gianni L, Bianchini G, Ali HR. Spatial predictors of immunotherapy response in triple-negative breast cancer. Nature. 2023 Sep;621(7980):868-876. doi: 10.1038/s41586-023-06498-3. Epub 2023 Sep 6. PMID 37674077